CLINICAL TRIAL: NCT00247390
Title: A Randomised, Double-blind, Placebo-controlled Study to Determine the Long-term Efficacy and Safety of Ramelteon in Adults With Chronic Insomnia.
Brief Title: Long-Term Efficacy and Safety of Ramelteon in Adults With Chronic Insomnia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: VP, Clinical Science, Takeda Global Research & Development Centre (Europe) Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-375-EC302; 2004-004351-20; U1111-1114-3231 (Registry Identifier: WHO)
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Insomnia
Keywords: Chronic Insomnia; Sleep Initiation and Maintenance Disorder; Drug Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramelteon 8 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 8 mg, tablets, orally, once daily for up to 42 weeks.
  Other Names: Rozerem; TAK-375
  Arms: Ramelteon 8 mg QD
Drug: Placebo — Ramelteon placebo-matching tablets, orally, once daily for up to 42 weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of this study to determine the long-term efficacy and safety of ramelteon, once daily (QD).

DETAILED DESCRIPTION:
A vast majority of people are affected by chronic insomnia in the western world. Several studies have looked at this and have estimated that 30% to 48% of the general population is affected at some time in their life with a form of insomnia that goes on for several months, and about one third of those are described as severely affected. Daytime symptoms of insomnia include tiredness, lack of energy, difficulty concentrating, and irritability. Recent epidemiologic research focusing on the quality of life has identified significant insomnia-related conditions that relate to work productivity, health care utilization, and risk of depression. Insomnia is associated with diminished work output, absenteeism, and greater rates of accidents.

An ideal treatment for chronic insomnia would include administration of therapy for an extended period. Specifically, it should be safe and effective for a period longer than the 7 to 10 days to which use of the current drugs approved for short-term use are limited.

Because of the absence of evidence of residual effects in pre-clinical studies and phase 2 and 3 clinical trials, ramelteon may be a candidate for extended use. As chronic insomnia becomes more prevalent, there is a need to assess the long-term efficacy and safety of nightly dosing with ramelteon in the general population. Study participation is anticipated to be about 8 months and 3 weeks.

ELIGIBILITY:
Inclusion Criteria

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Body mass index between 18 and 34, inclusive.
* Based on sleep history, has had chronic insomnia for at least 3 months.
* Based on sleep history, reports a subjective sleep latency greater than or equal to 45 min and a subjective total sleep time less than or equal to 6.5 hours.
* Based on sleep history, habitual bedtime is between 10:00 PM and 1:00 AM.
* Mean latency to persistent sleep of greater than 20 minutes on two consecutive screening nights with neither night less than 15 minutes. Also, a mean of 60 minutes of wake time during the 480 minutes in bed across two nights with no night less than 45 minutes.
* Based on sleep history, normally uses pharmacological assistance to sleep 0 to 4 times per week in the last 3 months.

Exclusion Criteria

* Known hypersensitivity to ramelteon or related compounds, including melatonin, and melatonin related compounds.
* Participated in any other investigational study and/or taken any investigational drug within 30 days or five half-lives prior to the first dose of single-blind study medication, whichever is longer.
* Sleep schedule changes required by employment (eg, shift worker) within three months prior to the administration of single-blind study medication.
* Flown across greater than three time zones within 7 days prior to or during screening.
* Participated in a weight loss program or has substantially altered their exercise routine within 30 days prior to the administration of single-blind study medication.
* Has ever had a history of seizures, sleep apnea, restless leg syndrome, periodic leg movement syndrome, chronic obstructive pulmonary disease or fibromyalgia.
* History of psychiatric disorder within the past 6 months.
* History of alcohol abuse within the past 12 months, as defined in Diagnostic & Statistical Manual of Mental Disorders, 4th Edition Revised, or regularly consumes more than 14 alcoholic drinks per week, or consumed any alcoholic drinks within 24 hours of any polysomnogram visits.
* History of drug abuse within the past 12 months, as defined in Diagnostic & Statistical Manual of Mental Disorders, 4th Edition Revised.
* Current significant hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematologic, neurological, or metabolic disease, unless currently controlled and stable with protocol-allowed medication, within 30 days prior to the first night of single-blind study medication.
* Apnea hypopnea index (per hour of sleep) greater than 10 as seen on the first polysomnogram screening night.
* Periodic Leg Movement Syndrome with arousal index (per hour of sleep) greater than 10 as seen on the first polysomnogram screening night.
* Positive urine drug screen at Screening Visit 1 or any of the polysomnogram assessment visits.
* Positive breathalyzer test on any of the polysomnogram assessment visits.
* Uses tobacco products (including nicotine gum and patch) or any other products that may interfere with the sleep wake cycle during nightly awakenings.
* Used any central nervous system medication or other drugs or supplements known to affect sleep/wake function within 1 week (or 5 half lives of the drug, whichever is longer) prior to the administration of single-blind study medication. These medications must not have been used to treat psychiatric disorders.
* Intends to continue taking any disallowed medication or any prescription medication or over the counter medication that is known to affect the sleep/wake function or otherwise interfere with evaluation of the study medication. The subject must report all prescription and over the counter medications taken in the three weeks prior to screening.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Anxiolytics
  * Sedatives
  * Hypnotics
  * CNS active drugs (including herbal)
  * Antidepressants
  * Narcotic analgesics
  * Anticonvulsants
  * Beta blockers
  * Sedating H1 antihistamines
  * St. John's Wort
  * Systemic steroids
  * Kava-kava
  * Respiratory stimulants
  * Ginkgo-biloba
  * Decongestants
  * Over-the-counter and prescription stimulants
  * Antipsychotics
  * Over-the-counter and prescription diet aids
  * Muscle Relaxants
  * Melatonin and all other drugs or supplements known to affect sleep/wake function
* Any additional condition(s) that in the Investigator's opinion would

  * affect sleep/wake function
  * prohibit the subject from completing the study
  * indicate that continuation in the study would not be in the best interests of the subject.
* History of hepatitis B or hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2005-07; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Mean change in Latency to Persistent Sleep of 2-night polysomnogram. | Months 3 and 6 or Final Visit

SECONDARY OUTCOMES:
Mean change in Total Sleep Time from polysomnogram, on 2 nights over 6 months. | Week 1 and Months 1, 3, 5 and 6 or Final Visit
Mean change in Subjective Sleep Latency by postsleep questionnaire on 2 nights over 6 months. | Week 1 and Months 1, 3, 5 and 6 or Final Visit
Mean change in Subjective Total Sleep Time by postsleep questionnaire on 2 nights over 6 months. | Week 1 and Months 1, 3, 5 and 6 or Final Visit
Mean change in Subjective Number of Awakenings by postsleep questionnaire. | Week 1 and Months 1, 3, 5 and 6 or Final Visit
Mean change in Subjective Sleep Quality by postsleep questionnaire. | Week 1 and Months 1, 3, 5 and 6 or Final Visit
Total Sleep Time in rapid eye movement (REM) sleep as determined by polysomnogram. | Week 1 and Months 1, 3, 5 and 6 or Final Visit
Total Sleep Time in stage 1 non-rapid eye movement (NREM) sleep as determined by polysomnogram. | Week 1 and Months 1, 3, 5 and 6 or Final Visit
Total Sleep Time in stage 2 non-rapid eye movement (NREM) sleep as determined by polysomnogram. | Week 1 and Months 1, 3, 5 and 6 or Final Visit
Total Sleep Time in stage 3/4 non-rapid eye movement (NREM) sleep as determined by polysomnogram. | Week 1 and Months 1, 3, 5 and 6 or Final Visit
Total Sleep Time in stage 1 sleep as determined by polysomnogram. | Week 1 and Months 1, 3, 5 and 6 or Final Visit
Latency to Rapid Eye Movement as determined by polysomnogram. | Week 1 and Months 1, 3, 5 and 6 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (48):
- United States (19):
  - Birmingham, Alabama
  - Hot Springs, Arkansas
  - Los Angeles, California
  - Oakland, California
  - San Diego, California
  - Santa Monica, California
  - Miami, Florida
  - Naples, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Overland Park, Kansas
  - Louisville, Kentucky
  - Chevy Chase, Maryland
  - Lincoln, Nebraska
  - New York, New York
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Columbia, South Carolina
  - Austin, Texas
- Australia (4):
  - Adelaide
  - Camperdown
  - Melbourne
  - Victoria
- Belgium (2):
  - Brussels
  - Edegem
- Czechia (3):
  - České Budějovice
  - Ostrava-Poruba
  - Prague
- Finland (3):
  - Espoo
  - Helsinki
  - Turku
- France (5):
  - Bron
  - Clamart
  - Garches
  - Paris
  - Rouffach
- Germany (6):
  - Berlin
  - Göttingen
  - Hamburg
  - Münster
  - Schwalmstadt
  - Schwerin
- Milan, Italy
- Russia (5):
  - Irkutsk
  - Moscow
  - Saint Petersburg
  - Samara
  - Yekateringburg

REFERENCES:
- [Result] Mayer G, Wang-Weigand S, Roth-Schechter B, Lehmann R, Staner C, Partinen M. Efficacy and safety of 6-month nightly ramelteon administration in adults with chronic primary insomnia. Sleep. 2009 Mar;32(3):351-60. doi: 10.1093/sleep/32.3.351. PMID 19294955
- [Result] Wang-Weigand S, McCue M, Ogrinc F, Mini L. Effects of ramelteon 8 mg on objective sleep latency in adults with chronic insomnia on nights 1 and 2: pooled analysis. Curr Med Res Opin. 2009 May;25(5):1209-13. doi: 10.1185/03007990902858527. PMID 19327100
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI